CLINICAL TRIAL: NCT00741962
Title: A Pilot Double-Blind Crossover Study on the Effects of VR-3 Herbal Blend Intake on Acute and Chronic Stress and Their Biomarkers in Healthy Adults
Brief Title: A Study on the Effects of VR-3 Herbal Blend Intake on Acute and Chronic Stress in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NEMA Research, Inc. (Industry)
Responsible Party: Dr. Ismail Shalaby, CEO, NEMA Research, Inc.,
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Adaptogen Study 001
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: VR-3 Herbal Blend
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: VR-3 Herbal Blend — This is a liquid blend of various reputed adaptogenic herbs. The dosage will be 2ml of liquid per day.
  Arms: 1
Dietary Supplement: Placebo — The placebo will be a similar tasting liquid as VR-3 Herbal blend. The dosage will be 2ml of liquid per day.
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of VR-3 Herbal Blend and its effects on acute and chronic stress responses.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 35-45
2. No health concerns as determined by study physicians
3. Women must not be pregnant or become pregnant for the duration of the study.

Exclusion Criteria:

1. The subject has a history of hypersensitivity to any of the compounds used in the study
2. The subject is pregnant or a lactating female. Note: If the potential subject is a post-menarcheal female, a pregnancy test (urine or serum) must be performed within 24 hours of study drug administration and confirmed negative in order for the potential subject to be enrolled).
3. History of Psychiatric Illness or Chronic Stress or Anxiety
4. Hypertension, cardiovascular disease, or other health concerns that may confound study results
5. Allergy or sensitivity to test product or ingredients
6. Individuals who are cognitively impaired or who are not able to give informed consent
7. Clinically significant or abnormal laboratory result that can confound the study
8. Medication or nutraceutical intake that can interact with the adaptogens or the biomarkers used in the study (to be determined by study physician)
9. Previous participation in a clinical research trial within 30 days prior to randomization
10. The subject has an ongoing abuse of illicit substances, alcohol, or actively smoking marijuana.
11. The subject is actively engaging in the use of Herbal Medicine, Traditional Chinese Medicine, Ancient Indian Medicine, Yoga, or Ayurveda

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change in salivary alpha-amylase and cortisol as stress biomarkers for the acute and chronic stress response following VR-3 Herbal Blend use | 10 weeks

SECONDARY OUTCOMES:
Change in acute psychological stress | 10 weeks
Change in chronic stress | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- NEMA Research, Naples, Florida, United States